CLINICAL TRIAL: NCT02782819
Title: A Randomized Controlled Trial of Crystalloid Alone Versus Crystalloid Plus Colloid in Shock Resuscitation
Brief Title: A Comparison of Crystalloid Alone Versus Crystalloid Plus Colloid in Shock Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Surat Tongyoo, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si685/2014
Record Dates: First submitted 2016-05-16; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Hypotension and Shock
Keywords: Shock resuscitation; colloid; crystalloid
MeSH Terms: conditions — Hypotension; Shock | interventions — Crystalloid Solutions; Colloids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crystalloid (Placebo Comparator): Isotonic crystalloid solution resuscitation
  Interventions: Drug: Isotonic crystalloid solution resuscitation
- Crystalloid plus Colloid (Active Comparator): Colloid solution resuscitation
  Interventions: Drug: Isotonic crystalloid solution resuscitation; Drug: Colloid solution resuscitation

INTERVENTIONS:
Drug: Isotonic crystalloid solution resuscitation — Patient will receive normal saline or Ringer lactate or other balance salt solution during fluid resuscitation for shock reversal.
  Other Names: Crystalloid
Drug: Colloid solution resuscitation — Patient will receive 5% albumin or gelatin solution during shock resuscitation
  Other Names: Colloid plus
  Arms: Crystalloid plus Colloid

SUMMARY:
Fluid resuscitation is the most effective treatment of shock. Isotonic crystalloid solution is the current recommended initial fluid resuscitation. However, this kind of fluid has high volume of distribution and may require large volume administration before achieve therapeutic goal of shock reversal. There are rising concern about the delay in shock reversal and adverse consequences of large amount volume of fluid therapy. Colloid fluid have been used as the alternate fluid resuscitation, aiming to limit the volume of fluid resuscitation and promote shock reversal. Whether colloid infusion can improve shock reversal rate and decrease complication associated with fluid resuscitation, had inconclusive information.

DETAILED DESCRIPTION:
Fluid resuscitation is the most effective treatment of shock. Isotonic crystalloid solution is the current recommended initial fluid resuscitation. However, this kind of fluid has high volume of distribution and may require large volume administration before achieve therapeutic goal of shock reversal. There are rising concern about the delay in shock reversal and adverse consequences of large amount volume of fluid therapy. Colloid fluid have been used as the alternate fluid resuscitation, aiming to limit the volume of fluid resuscitation and promote shock reversal. Data from a recent randomized controlled study showed the improve long term survival among shock patients whose resuscitated with colloid solution. There were evidence about the increase incidence of acute kidney injury among critically ill patients who received hydroxyethyl starch, a previously worldwide used colloid solution. For septic shock, the leading cause of shock in current situation, resuscitation with albumin may associated with better outcome, while increasing mortality had been reported among the patient who received hydroxyethyl starch. Whether colloid infusion can improve shock reversal rate and decrease complication associated with fluid resuscitation, had inconclusive information.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* New onset of shock within 24 hours
* Mean arterial blood pressure less than 65 mmHg or systolic blood pressure less than 60% of patient's baseline blood pressure
* Evidence of poor tissue perfusion including: urine output less than 0.5 mL/kg/hr, lactate more than 2 mmol/L, alteration of consciousness without other explanation
* Evidence of fluid inadequacy (CVP < 12 mmHg, Pulmonary capillary wedge pressure < 18 mmHg) or evidence of fluid responsive (IVC diameter variation > 15%, pulse pressure variation > 15%, positive fluid challenge test)

Exclusion Criteria:

* Prolong shock more than 24 hours
* Received colloid solution more than 1,000 mL in previous 72 hours
* Do not resuscitation documented patient
* Contraindication for fluid therapy including: suspected cardiogenic shock, evidence of pulmonary edema, history of anaphylaxis after fluid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who had shock reversal | 6 hours after initial resuscitation
  Shock reversal was defined by mean arterial blood pressure > 65 mmHg plus lactate clearance more than 10%

SECONDARY OUTCOMES:
Mortality rate | 28 days
  Dead from any causes within 28 days after enrollment
Hospital mortality | 90 days
  Dead from any causes during hospital admission
Total fluid resuscitation within 24 hours | 24 hours
  Total volume of fluid resuscitation the patient received within 24 hours after enrollment
Renal replacement therapy | 28 days
  Patient who required acute renal replacement therapy during admission

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Permpikul, MD., Study Director — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Background] Annane D, Siami S, Jaber S, Martin C, Elatrous S, Declere AD, Preiser JC, Outin H, Troche G, Charpentier C, Trouillet JL, Kimmoun A, Forceville X, Darmon M, Lesur O, Reignier J, Abroug F, Berger P, Clec'h C, Cousson J, Thibault L, Chevret S; CRISTAL Investigators. Effects of fluid resuscitation with colloids vs crystalloids on mortality in critically ill patients presenting with hypovolemic shock: the CRISTAL randomized trial. JAMA. 2013 Nov 6;310(17):1809-17. doi: 10.1001/jama.2013.280502. PMID 24108515